CLINICAL TRIAL: NCT03131921
Title: Resting Energy Expenditure in Cancer - Associations With Body Composition, Dietary Intake, and Exercise Habits
Brief Title: Determining Energy Needs in Colorectal Cancer
Acronym: RECODE
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: HREBA.CC.15-0204; No grant number. (Other: National Institutes of Health)
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
Keywords: Energy expenditure; Nutrition; Colorectal cancer; Dietary needs
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Colorectal cancer: No intervention. Patients with newly diagnosed stage II-IV colorectal cancer will be enrolled.

SUMMARY:
This is an observational study to assess the determinants of energy expenditure in cancer, and how those change throughout the disease trajectory. The investigators hypothesize that skeletal muscle will be the primary determinant of energy expenditure throughout the disease trajectory.

DETAILED DESCRIPTION:
Proper nutrition is a hallmark of successful cancer treatment. Adequate energy intake helps to maintain body weight and composition, improving outcomes such as response to therapy, quality of life, and survival. Unfortunately, little is known about energy needs in cancer, as few studies have assessed energy expenditure (the amount of calories used/day). Furthermore, individuals with cancer often experience muscle loss (sarcopenia), changes in physical activity, and undergo treatment, all of which might substantially alter energy needs. Equations to estimate energy REE (and thus dietary requirements) were created from cohorts of healthy individuals, and no tools that can be easily used in clinical settings are validated to assess REE.

The overarching aim of this study is to evaluate the largest component of energy needs - resting energy expenditure (REE) in relation to body composition (skeletal muscle, adipose tissue) and physical activity in a cohort of patients with colorectal cancer. Other aims will explore the changes in energy expenditure and determine the accuracy of a portable indirect calorimeter for measuring REE.

Newly-diagnosed individuals with stage II-IV colorectal cancer will undergo indirect calorimetry to assess REE. Body composition will be measured by CT scans, with sarcopenia status based on previously published cut-points. Nutritional status and inflammation (C-reactive protein, neutrophil:lymphocyte) will be assessed as confounding variables.

Total energy expenditure will be measured near treatment start in a sub-sample of 20 participants with colorectal cancer using doubly labeled water and accelerometers. Participants will wear accelerometers (ActiCal) for 14 days to provide detailed physical activity data.These assessments will also be preformed in a sub-sample of 20 participants after treatment end.

An additional part of this study will assess the validity of a portable indirect calorimeter for measuring REE. To address this, a sub-group of patients will be invited to undergo an additional test of REE using a portable indirect calorimeter, the FitMate (COSMED). Results will be compared using Pearson's correlation, dependent samples t-test, and Bland-Altman analysis to assess agreement between the FitMate and validated indirect calorimeters (VMax metabolic cart and whole body calorimtery unit). Exploratory outcomes include phase angle by bioelectrical impedance analysis, handgrip strength, calf circumference, and nutrition status by patient generated subjective global assessment (PG-SGA).

The results from this project will provide a basis of better energy recommendations to sustain body weight and composition, thereby improving prognosis in cancer.

ELIGIBILITY:
Pre-treatment Participants:

Inclusion Criteria:

* Recent diagnosis of colorectal cancer (stage II-IV);
* Able to arrive at the Human Nutrition Research Unit fasted;
* Patients undergoing treatment should be able to undergo measurements within 20 days of treatment commencement;
* Able to provide written informed consent;
* Able to communicate freely in English;
* Age 18-90

Exclusion Criteria:

* Recent (within the past month) anti-cancer therapy;
* Recent invasive surgery (within the last 4 weeks);
* Women during pregnancy or are breast-feeding;
* Inability to breathe under the indirect calorimeter hood for 20-30 minutes;
* Severe toxicity during the 1st cycle therapy (where applicable);
* Severe mobility issues (e.g. confined to wheelchair);
* Use of medications that may affect body composition or metabolism will be evaluated individually (e.g. cortico-steroids, hormone replacement, etc.)
* Patients with a pacemaker

Post-treatment participants:

Inclusion Criteria

* Recently (<3 year) completed adjuvant chemotherapy treatment for colorectal cancer (stage II-IV)
* Able to arrive at the Human Nutrition Research Unit fasted
* Able to provide written informed consent
* Able to communicate freely in English
* Age 18-90

Exclusion Criteria

* Recent (within the past month) anti-cancer therapy
* Recent invasive surgery (within the last 4 weeks)
* Women during pregnancy or are breast-feeding
* Inability to breathe under the indirect calorimeter hood for 20-30 minutes
* Severe mobility issues (e.g. confined to wheelchair)
* Use of medications that may affect body composition or metabolism will be evaluated individually (e.g. cortico-steroids, hormone replacement, etc.)
* Patients with a pacemaker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer (stage II-IV) at the Cross Cancer Institute (Edmonton, Alberta, Canada)
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Resting energy expenditure | At baseline, before or immediately beginning cancer treatment
  To assess resting energy expenditure using indirect calorimtery

SECONDARY OUTCOMES:
Body composition | At baseline, before or immediately beginning cancer treatment
  To assess skeletal muscle and adipose tissue using computerized tomography images taken before beginning cancer treatment
Total energy expenditure | Post-treatment, within 3 years after completion of cancer treatment
  To assess total energy expenditure (one time, over 14 days) using doubly labeled water and accelerometers

CONTACTS AND LOCATIONS:
Overall Officials: Carla M Prado, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Cross Cancer Institute, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prado CM, Lieffers JR, McCargar LJ, Reiman T, Sawyer MB, Martin L, Baracos VE. Prevalence and clinical implications of sarcopenic obesity in patients with solid tumours of the respiratory and gastrointestinal tracts: a population-based study. Lancet Oncol. 2008 Jul;9(7):629-35. doi: 10.1016/S1470-2045(08)70153-0. Epub 2008 Jun 6. PMID 18539529
- [Background] Purcell SA, Elliott SA, Baracos VE, Chu QS, Prado CM. Key determinants of energy expenditure in cancer and implications for clinical practice. Eur J Clin Nutr. 2016 Nov;70(11):1230-1238. doi: 10.1038/ejcn.2016.96. Epub 2016 Jun 8. PMID 27273068
- [Background] Moses AW, Slater C, Preston T, Barber MD, Fearon KC. Reduced total energy expenditure and physical activity in cachectic patients with pancreatic cancer can be modulated by an energy and protein dense oral supplement enriched with n-3 fatty acids. Br J Cancer. 2004 Mar 8;90(5):996-1002. doi: 10.1038/sj.bjc.6601620. PMID 14997196
- [Background] Skipworth RJ, Stene GB, Dahele M, Hendry PO, Small AC, Blum D, Kaasa S, Trottenberg P, Radbruch L, Strasser F, Preston T, Fearon KC, Helbostad JL; European Palliative Care Research Collaborative (EPCRC). Patient-focused endpoints in advanced cancer: criterion-based validation of accelerometer-based activity monitoring. Clin Nutr. 2011 Dec;30(6):812-21. doi: 10.1016/j.clnu.2011.05.010. Epub 2011 Jul 5. PMID 21733604
- [Background] Reeves MM, Battistutta D, Capra S, Bauer J, Davies PS. Resting energy expenditure in patients with solid tumors undergoing anticancer therapy. Nutrition. 2006 Jun;22(6):609-15. doi: 10.1016/j.nut.2006.03.006. PMID 16704954
- [Background] Kyle UG, Soundar EP, Genton L, Pichard C. Can phase angle determined by bioelectrical impedance analysis assess nutritional risk? A comparison between healthy and hospitalized subjects. Clin Nutr. 2012 Dec;31(6):875-81. doi: 10.1016/j.clnu.2012.04.002. Epub 2012 May 4. PMID 22560739
- [Derived] Purcell SA, Elliott SA, Walter PJ, Preston T, Cai H, Skipworth RJE, Sawyer MB, Prado CM. Total energy expenditure in patients with colorectal cancer: associations with body composition, physical activity, and energy recommendations. Am J Clin Nutr. 2019 Aug 1;110(2):367-376. doi: 10.1093/ajcn/nqz112. PMID 31225583